CLINICAL TRIAL: NCT06101680
Title: RhabdomYolyse in Intensive caRe
Acronym: RYR
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Arnaud WIEDEMANN-FODE, Clinical Professor, Central Hospital, Nancy, France
Other Study IDs: 2022PI201
Record Dates: First submitted 2023-10-16; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Rhabdomyolysis
Keywords: rhabdomyolysis; child; Intensive Care
MeSH Terms: conditions — Rhabdomyolysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children in intensive care with rhabdomyosis

SUMMARY:
Analysis of the outcome of patients < 18 years old, treated in an intensive care unit for severe rhabdomyolysis, regardless of etiology (renal failure rate, death rate, organ replacement rate)

ELIGIBILITY:
Inclusion Criteria:

* CPK > 5000 UI/L
* Care in Pediatric Intensive Care Unit
* Age < 18 years old

Exclusion Criteria:

* Parental refusal

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with severe rhabdomyolysis (> 5000 UI/L) hospitalized in intensive care unit.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Use of renal remplacement therapy | 7 days after admission in intensive care unit
  Use of renal remplacement therapy in case of severe rhabdomyolysis in children in intensive care unit

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Wiedemann, MD PhD, Principal Investigator — CHRU Nancy
Locations (1):
- Reanimation Pediatrique, Nancy, France